CLINICAL TRIAL: NCT04646577
Title: The Effect of Transcranial Direct Current Stimulation Combined With Functional Task Training on Motor Recovery in Stroke Patients
Brief Title: The Effect of tDCS Combined With Functional Task Training on Motor Recovery in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Fahad Specialist Hospital Dammam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NEU0329
Record Dates: First submitted 2020-10-06; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Stroke; Stroke, Acute; Motor Function
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Device: Transcranial Direct Current Stimulation (tDCS
- Sham (Sham Comparator)
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Subjects will either undergo (1) active low-frequency rTMS (1Hz continuous) prime with anodal Transcranial Direct Current Stimulation (tDCS) on the affected side combine with Constraint induced movement therapy. Each session will last 20 minutes.
  Arms: Active
Device: Transcranial Direct Current Stimulation (tDCS — Subjects will either undergo sham Transcranial Direct Current Stimulation (tDCS) on the affected side combine with Constraint-induced movement therapy.

SUMMARY:
We propose to enhance the effects of brain plasticity using a powerful noninvasive technique for brain modulation consisting of navigated transcranial magnetic stimulation (TMS) priming with transcranial direct current stimulation (tDCS) in combination with motor-training-like constraint-induced movement therapy (CIMT).

ELIGIBILITY:
Inclusion Criteria:

1. age 18-90
2. first-time clinical ischemic or hemorrhagic cerebrovascular accident as noted in the radiological (or physician's) report;
3. the ability to extend =20° at the wrist and 10° at the metacarpophalangeal and interphalangeal joints of all digits;
4. participants must demonstrate adequate balance while wearing the restraint;
5. the ability to stand from a sitting position and the ability to stand for at least 2 minutes with or without upper extremity support;
6. weakness, defined as score of 15-55 (out of 66) on arm motor Fugl-Meyer (FM) scale; and
7. stroke onset more then 6 months prior to study enrollment.

Exclusion Criteria:

1. significant pre-stroke disability;
2. where applicable (a history of depression before the stroke);
3. any substantial decrease in alertness, language reception, or attention that might interfere with understanding the instructions for the motor testing;
4. excessive pain in any joint of the paretic extremity;
5. contraindications to single-pulse TMS (TMS will be used to measure cortical excitability) such as metal head implants;
6. advanced liver, kidney, cardiac, or pulmonary disease;
7. a terminal medical diagnosis consistent with survival 1 year;
8. coexistent major neurological or psychiatric disease (to decrease the number of confounders);
9. a history of significant drug abuse in the prior 6 months;
10. the use of certain neuropsychotropic drugs such as tricyclics, antidepressants, or 51 of 66 carbamazepine;
11. active enrollment in a separate intervention study targeting stroke recovery; (
12. previously applied constraint-induced motor therapy and/or tDCS treatment for stroke; and
13. a history of epilepsy before stroke (or episodes of seizures within the last six months).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
To assess the neurophysiologic findings of cortical plasticity. | Before 10 sessions, before and after each session (every day), after 10 daily sessions and after 6 weeks
  Expressed as percent motor resting threshold and numerical values of motor evoked potential. The motor evoked potential (MEP) will be provided by twenty unconditioned stimuli (120% of motor resting threshould). The percentage of inhibition or facilitation for each before and after stimulation will be calculated.
To assess the motor function changes . | before 10 sessions, before and after each session (every day), after 10 daily sessions and after 30 days
  Change from motor hand function: ordinal variable measured through the Jebsen-Taylor Hand Function Test (JTHFT). The JTHFT has seven subsets which are writing, simulated page-turning, lifting small objects, simulated feeding, stacking, and lifting large, lightweight, and heavy objects

SECONDARY OUTCOMES:
Sensory-motor function of the upper limb | before 10 sessions, before and after each session (every day), after 10 daily sessions and after 30 days
  This consists of a quantitative scale developed to measure (motor recovery, balance, sensation, and some joint function) recovery of the motor function of stroke patients. Measured through the Fugl-Meyer Rating Scale, which expressed in values from 0 to 66.
Degree of disability: | before 10 sessions, before and after each session (every day), after 10 daily sessions and after 30 days
  This consists of a quantitative scale developed to measured the disability caused by impairments in stroke patients. The Barthel Index Score (Activities of Daily Living) measured through ranges from 0 to 20, principally concerned with physical aspects of disability.

REFERENCES:
- [Derived] Al-Hussain F, Nasim E, Iqbal M, Altwaijri N, Asim N, Yoo WK, Bashir S. The effect of transcranial direct current stimulation combined with functional task training on motor recovery in stroke patients. Medicine (Baltimore). 2021 Feb 12;100(6):e24718. doi: 10.1097/MD.0000000000024718. PMID 33578615